CLINICAL TRIAL: NCT03158402
Title: High Intensity Preoperative Inspiratory Muscle Training (IMTHi) Effects on the Perioperative Inflammatory Reaction in Cardiac Surgery With an Associated Biocollection.
Brief Title: Preoperative Inspiratory Muscle Training Effects on the Perioperative Inflammatory Reaction in Cardiac Surgery.
Acronym: EMI HiPo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-A00216-47
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Thoracic Surgery; Prehabilitation; Respiratory Therapy
Keywords: Inspiratory muscle training; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham IMT (Sham Comparator): Preoperative Inspiratory muscle training at low intensity (15% Pimax) which is considered as a no effect training.
  Interventions: Other: Prehabilitation with inspiratory muscle training
- Hi Intensity IMT (Experimental): High intensity muscle training in the preoperative period at 80% of the maximal inspiratory muscle pressure.
  Interventions: Other: Prehabilitation with inspiratory muscle training

INTERVENTIONS:
Other: Prehabilitation with inspiratory muscle training — 3 to 6 weeks of two times a day inspiratory muscle training at 80% of the Maximum Inspiratory Pressure.

SUMMARY:
This study evaluates the impact of preoperative high-intensity inspiratory muscle training (IMThi) before cardiac surgery on perioperative inflammatory response. Half participants will receive high intensity inspiratory muscle training and the others a sham inspiratory muscle therapy.

ELIGIBILITY:
Inclusion Criteria:

* Waiting for thoracic surgery with valve replacement
* Preoperative surgeon consultation between 3 and 6 weeks before surgery

Exclusion Criteria:

* Patient with antecedent of lung surgery
* Patient with neuromuscular or neurovascular disease
* Non anticipated surgery with a time between surgeon consultation and surgery inferior to 3 weeks.
* Inhability to do the preoperative exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Preoperative STNFr1 level | Outcome is evaluated at the training initiation and re evaluated 24hours before the surgery
  Post training and preoperative Serum concentration of the SRNFr1 cytokine.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Angers, Angers, France

REFERENCES:
- [Result] Furon Y, Dang Van S, Blanchard S, Saulnier P, Baufreton C. Effects of high-intensity inspiratory muscle training on systemic inflammatory response in cardiac surgery - A randomized clinical trial. Physiother Theory Pract. 2024 Apr;40(4):778-788. doi: 10.1080/09593985.2022.2163212. Epub 2023 Jan 13. PMID 36637368